CLINICAL TRIAL: NCT03047070
Title: Lidocaine Infusion in Functional Endoscopic Sinus Surgery
Brief Title: Lidocaine in ERAS for FESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SM22017
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): IV Lidocaine infusion
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): IV normal saline infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — IV Lidocaine infusion
  Arms: Lidocaine
Drug: Normal saline — IV normal saline infusion
  Arms: Control

SUMMARY:
Functional endoscopic sinus surgery (FESS) is a commonly performed procedure. It is known that bleeding during FESS can affect directly to the visibility of safe landmarks and surgical outcomes.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a commonly performed procedure in the head and neck field. It is known that bleeding during FESS can affect directly to the visibility of safe landmarks and surgical outcomes.

Use of vasoactive drugs to control bleeding is not without pitfalls. Systemic effects of epinephrine may constitute a potential hazard in patients with hypertension, ischemic heart disease, anemia, preexistent liver or renal damage and endocrine dysfunction (hyperthyroidism, pheochromocytoma and diabetes mellitus).

Lidocaine is a prototypical local anesthetic, but it also has systemic effects that are mediated by inhibitory effects on N-methyl-d-aspartate receptors and leukocyte priming. Consequently, systemic lidocaine is antiinflammatory, analgesic, and antihyperalgesic. Randomized clinical trials, however, have produced mixed results. Several studies have shown reduction in postoperative opioid consumption and pain scores, whereas others have failed to show a benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 20-50 yr ASA class I and II
* Elective Functional endoscopic sinus surgery (FESS) under general anesthesia.

Exclusion Criteria:

* Patient refusal, allergy to the study medication, pre-existing chronic pain at any site requiring treatment, intolerance to nonsteroidal anti-inflammatory drugs (NSAIDs), psychiatric or neurological disorders, seizure disorder requiring medication within the previous 2 years, body mass index > 30 kg/ m2, revision sinus surgery, pregnancy, and patients with cardiovascular, cerebrovascular, respiratory, renal or hepatic diseases

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding | Intraoperative assessment till end of operation
  Will be calculated from the fluid volume of the suction canister. The volume of irrigating fluid will subtracted from the total volume of fluid contained in the suction bottle. Additionally, a fully soaked cotton strip will be assumed to contain 5 ml of blood and a partially soaked one to contain 2-3 ml of blood

SECONDARY OUTCOMES:
Quality of surgical field | intraoperative assessment
  The surgeon will assess the quality of surgical field every 15 min after the beginning of drug infusion for the first 60 min according to a 6-point Boezaart scale
Surgeon satisfaction | At the end of surgery
  with a 4-point scale: 1 = Poor, 2 = Moderate, 3 = Good, 4 = Excellent
Mean arterial pressure | intraoperative assessment
  Will be assessed at the initial phase (baseline), immediately after induction of anesthesia, and then 15, 30. 45, 60 min after the begining of drug infusion
Heart rate | intraoperative assessment
  Will be assessed at the initial phase (baseline), immediately after induction of anesthesia, and then 15, 30. 45, 60 min after the begining of drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Faculty of Medicine Assuit University, Asyut, Assuit
  - Seham Mohamed Moeen Ibrahim, Asyut

IPD SHARING:
Plan to Share IPD: No